CLINICAL TRIAL: NCT01044264
Title: A Randomized, Double-Blind, Multiple-Site, Placebo-Controlled Study Comparing Two 1% Clindamycin/5% Benzoyl Peroxide Topical Gel Formulations in the Treatment of Moderate to Severe Acne Vulgaris
Brief Title: Clinical Study Between Two 1% Clindamycin/5% Benzoyl Peroxide Topical Gel Formulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAC-501-601-727998; NCT00807638 (obsolete NCT alias)
Record Dates: First submitted 2010-01-04; First posted 2010-01-07 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; bioequivalency; clindamycin; benzoyl peroxide
MeSH Terms: conditions — Acne Vulgaris | interventions — clindamycin phosphate benzoyl peroxide combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1% Clindamycin/5% Benzoyl Peroxide Topical Gel (Active Comparator): Test product
  Interventions: Drug: 1% Clindamycin/5% Benzoyl Peroxide Topical Gel
- DUAC® 1% Clindamycin/5% Benzoyl Peroxide Topical Gel (Active Comparator): Reference product
  Interventions: Drug: 1% Clindamycin/5% Benzoyl Peroxide Topical Gel
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1% Clindamycin/5% Benzoyl Peroxide Topical Gel — Topical Gel
  Other Names: DUAC® 1% Clindamycin/5% Benzoyl Peroxide Topical Gel
  Arms: 1% Clindamycin/5% Benzoyl Peroxide Topical Gel; DUAC® 1% Clindamycin/5% Benzoyl Peroxide Topical Gel
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A randomized, double-blind, multiple-site, placebo-controlled, parallel-group clinical study conducted to evaluate the bioequivalence of two 1% Clindamycin/5% Benzoyl Peroxide Topical Gel formulations.

ELIGIBILITY:
Inclusion Criteria:

* healthy men or women, 12 years of age and older
* willing to participate and sign a copy of the informed consent form
* moderate to severe facial acne

Exclusion Criteria:

* history of allergy or hypersensitivity to clindamycin or benzoyl peroxide
* pregnant or lactating women
* evidence of a clinically significant disorder
* receipt of any drugs as part of a research study within 30 days prior to study dosing
* use of systemic, topical or facial products which may interfere with study
* significant facial hair, tattoos, excessive facial scarring, active facial sunburn, or peeling due to sunburn

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 602 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: FIRST PATIENT ENROLLED: 12/11/2007 LAST PATIENT COMPLETED: 9/18/2008
Groups:
- 1% Clindamycin/5% Benzoyl Peroxide Topical Gel: Test product
  1% Clindamycin/5% Benzoyl Peroxide Topical Gel : Topical Gel
- DUAC® 1% Clindamycin/5% Benzoyl Peroxide Topical Gel: Reference product
  1% Clindamycin/5% Benzoyl Peroxide Topical Gel : Topical Gel
- Placebo: Placebo : Placebo
Period: Overall Study
Arm/Group | 1% Clindamycin/5% Benzoyl Peroxide Topical Gel | DUAC® 1% Clindamycin/5% Benzoyl Peroxide Topical Gel | Placebo
Started | 200 | 202 | 200
Completed | 110 | 108 | 108
Not Completed | 90 | 94 | 92

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% Clindamycin/5% Benzoyl Peroxide Topical Gel | DUAC® 1% Clindamycin/5% Benzoyl Peroxide Topical Gel | Placebo | Total
Number analyzed (Participants) | 200 | 202 | 200 | 602
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 117 | 113 | 113 | 343
  Between 18 and 65 years | 83 | 89 | 87 | 259
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.2 (7.3) | 19.5 (7.1) | 20.1 (8.3) | 19.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 101 | 113 | 317
  Male | 97 | 101 | 87 | 285
Region of Enrollment [Number; unit: participants]
  United States | 200 | 202 | 200 | 602

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Inflammatory Lesions
Description: The primary endpoint of the study was the mean percent reduction from baseline to week 11 in inflamed lesion count (papules and pustules).
Time Frame: Baseline and week 11
Population: per-protocol population
Measure: Number; unit: percentage reduction of lesions
Arm/Group | 1% Clindamycin/5% Benzoyl Peroxide Topical Gel | DUAC® 1% Clindamycin/5% Benzoyl Peroxide Topical Gel | Placebo
Number analyzed (Participants) | 110 | 108 | 185
percentage reduction of lesions | 64.39 | 63.10 | 49.89
Statistical Analysis 1: Comparison: 1% Clindamycin/5% Benzoyl Peroxide Topical Gel vs DUAC® 1% Clindamycin/5% Benzoyl Peroxide Topical Gel; Test type: Non-Inferiority or Equivalence — BE of the test to reference in the per protocol population; Wilcoxon Rank Sum Test; Wilcoxon Rank Sum Test = 100, 90% CI 2-sided [92.47 to 113.54]

ADVERSE EVENTS:
Time Frame: 11 week treatment period
Arm/Group | 1% Clindamycin/5% Benzoyl Peroxide Topical Gel | DUAC® 1% Clindamycin/5% Benzoyl Peroxide Topical Gel | Placebo
Serious Adverse Events (participants affected / at risk) | 1 | 0 | 1
Other Adverse Events (participants affected / at risk) | 40/200 | 35/202 | 28/200
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | 1% Clindamycin/5% Benzoyl Peroxide Topical Gel | DUAC® 1% Clindamycin/5% Benzoyl Peroxide Topical Gel | Placebo
Kidney Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/200 (1) | 0/202 (0) | 0/200 (0)
Hematuria (Renal and urinary disorders) | 1/200 (1) | 0/202 (0) | 0/200 (0)
Mild Bipolar Conduct Disorder (Psychiatric disorders) | 0/200 (0) | 0/202 (0) | 1/200 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1% Clindamycin/5% Benzoyl Peroxide Topical Gel (N=200) | DUAC® 1% Clindamycin/5% Benzoyl Peroxide Topical Gel (N=202) | Placebo (N=200)
application site dryness (Skin and subcutaneous tissue disorders) | 25 | 21 | 21
headache (Nervous system disorders) | 3 | 8 | 3
Nasopharyngitis (Ear and labyrinth disorders) | 4 | 3 | 2
Application Site Burning (Skin and subcutaneous tissue disorders) | 4 | 2 | 1
Influenza (Infections and infestations) | 4 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other